CLINICAL TRIAL: NCT06045585
Title: Early Exploratory Clinical Study of the Safety, Tolerability and Initial Efficacy of JY231 Injection in the Treatment of Relapsed or Refractory B-cell Lymphoma
Brief Title: JY231 Injection in the Treatment of Relapsed or Refractory B-cell Lymphoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Second Provincial General Hospital (Other)
Responsible Party: Principal Investigator, Qing Zhang, Chief Physician, Guangdong Second Provincial General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JY-CT-23-002
Record Dates: First submitted 2023-09-11; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Relapsed or Refractory B-cell Lymphoma
Keywords: JY231injection; Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell; Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- infusion of JY231 injection (Experimental): Infusion of JY231 Injection by dose of 1-10 x10^6 TU/kg、 1-5 x10^7 TU/kg、 5-10 x10^7 TU/kg Administration method: intravenous infusion、intraperitoneally infusion、Lymph node infusion； Subjects will be treated with Fludarabine and Cyclophosphamide before cell infusion（PI evaluation is required）.
  Interventions: Biological: infusion of JY231 injection

INTERVENTIONS:
Biological: infusion of JY231 injection — Infusion of JY231 Injection by dose of 1-10 x10^6 TU/kg、 1-5 x10^7 TU/kg、 5-10 x10^7 TU/kg Administration method: intravenous infusion、intraperitoneally infusion、Lymph node infusion； Subjects will be treated with Fludarabine and Cyclophosphamide before cell infusion（PI evaluation is required）.

SUMMARY:
Early exploratory clinical study of the safety, tolerability and initial efficacy of JY231 injection in the treatment of relapsed or refractory B-cell lymphoma

DETAILED DESCRIPTION:
This is a single-center, single-arm, open-treatment clinical study. In this study, approximately 10-20 adult and elderly patients with CD19-positive relapsed or refractory B-cell lymphoma will be enrolled for JY231 infusion therapy. The safety of JY231 was evaluated by observing adverse events after cell therapy. Evaluate the effectiveness of JY231 treatment compared to the results of the subjects' own previous standard treatment regimens or base data. Blood, bone marrow, and cerebrospinal fluid were collected before and 12 months after the JY231 infusion to detection.

ELIGIBILITY:
Inclusion Criteria:

1. understand and sign the informed consent and are willing and able to comply with all test requirements;
2. Age 18-75 years old, gender is not limited;
3. Flow cytometry or malignant tumor cells were CD19 positive;
4. Meet the clinical criteria for r/r B-cell lymphoma, including: indolent lymphoma (iNHL), follicular lymphoma (FL) and marginal zone lymphoma (MZL); Invasive B-cell lymphoma, including diffuse large B-cell lymphoma (DLBCL), primary mediastinal large B-cell lymphoma (PMBCL), transformed follicular lymphoma (TFL), and T-lymphocyt-rich large B-cell lymphoma (TCRBCL);
5. There is at least one measurable lesion on imaging (Lugano 2014 criteria), that is, a lymph node lesion with a diameter greater than 15 mm on CT cross-sectional images or an extranodal lesion with a diameter greater than 10 mm, with a positive FDG-PET test.
6. Expected survival ≥12 weeks;
7. The ECOG (Eastern Tumor Collaboration Group) score at baseline was 0 ~ 1;
8. Adequate organ function (indicators involving liver and kidney function can be appropriately relaxed) :

   * ALT ≤3 xULN;
   * AST)≤3x ULN;
   * Total bilirubin ≤1.5 x ULN;
   * Serum creatinine ≤ 1.5x ULN, or creatinine clearance ≥60 mL/min;
   * Indoor oxygen saturation ≥92%;
   * Left ventricular ejection fraction (LVEF) ≥55%, echocardiography confirmed no pericardial effusion, no clinically significant ECG findings;
   * No clinically significant pleural effusion;
9. Sufficient who with adequate bone marrow reserve, defined as:

   Absolute neutrophil count (ANC) > 1.000 /mm3; Absolute lymphocyte count (ALC) ≥300 /mm3; Platelet ≥50.000 /mm3; Hemoglobin > 8.0g/dl;
10. Using the following drugs must meet the following conditions:

    * Steroids: Therapeutic doses of steroids must be discontinued 72 hours before JY231 infusion. Physiological replacement doses of steroids are permitted;
    * Immunosuppression: Any immunosuppressive drug must be stopped ≥4 weeks prior to enrollment;
    * Anti-proliferative therapy other than lympho-depleting chemotherapy within two weeks of infusion; CD20 antibody therapy must be discontinued within 4 weeks prior to infusion or 5 half-lives (whichever is older);
    * CNS disease prevention must be stopped 1 week before JY231 infusion (e.g., intrathecal methotrexate).
11. Fertile men, to ensure that sexual partners can effectively prevent contraception; Women who are fertile, use effective birth control and consent to use birth control throughout the study period.

Exclusion Criteria:

1. Subjects with active cerebrospinal fluid malignant cells or brain metastases, or subjects with active central nervous system (CNS) lymphoma;
2. Subjects with a history of active CNS disease, such as seizures, cerebrovascular ischemia/bleeding, dementia, cerebellar disease, or any autoimmune disease involving the central nervous system;
3. Subjects who have received other study drugs within 30 days prior to screening;
4. Subjects who have previously received any anti-CD19 / anti-CD3 therapy or any other anti-CD19 therapy (except those with adequate bone marrow reserve and whose tumor is CD19-positive);
5. Patients who have previously been treated with any gene therapy product, including CAR-T therapy (except those with no CAR T in the body, normal T cell count and function, and CD19-positive tumors);
6. Subjects undergoing radiation therapy within 2 weeks prior to infusion;
7. Subjects with active hepatitis B (defined as hepatitis B virus DNA test value > 500 IU/mL) or hepatitis C (HCV RNA positive); Hiv-positive or treponem-positive subjects;
8. Subjects with an acute life-threatening bacterial, viral, or fungal infection that has not yet been controlled (e.g., positive blood culture ≤72 hours prior to infusion);
9. Participants with unstable angina pectoris and/or myocardial infarction in the 6 months prior to screening;
10. Subjects with prior or concurrent development of other malignancies, except in the following cases:

    * Adequately treated basal cell, thyroid papillary, squamous cell carcinomas (requiring adequate wound healing prior to enrollment);
    * Carcinoma in situ of cervical or breast cancer with curative treatment and no signs of recurrence for at least 3 years prior to the study;
    * The primary malignancy has been completely removed and in complete remission for ≥5 years.
11. Clinically significant ventricular arrhythmia;
12. Subjects received anticoagulant therapy within a week;
13. Active neuroautoimmune or inflammatory conditions (e.g. Guillian-Barre syndrome, amyotrophic lateral sclerosis);
14. Pregnant or lactating women, and female subjects who are planning to become pregnant within 2 years after JY231 injection infusion or male subjects whose partners plan to become pregnant within 2 years after JY231 injection infusion;
15. Subjects who, in accordance with the investigator's judgment and/or clinical standards, are contraindicated with any study procedure or have other medical conditions that may place them at unacceptable risk.
16. Other conditions that the investigator believes should not be included in this clinical trial, such as poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Month1、Month2、Month3、Month6、Month9、Month12
  Metric/method of measurement:IWG-2（2007）《Revised response criteria for malignant lymphoma》

CONTACTS AND LOCATIONS:
Overall Officials: Qing Zhang, Doctoral, Principal Investigator — Guangdong Second Provincial General Hospital
Locations (1):
- Guangdong Second Provincial General Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Pule MA, Straathof KC, Dotti G, Heslop HE, Rooney CM, Brenner MK. A chimeric T cell antigen receptor that augments cytokine release and supports clonal expansion of primary human T cells. Mol Ther. 2005 Nov;12(5):933-41. doi: 10.1016/j.ymthe.2005.04.016. Epub 2005 Jun 23. PMID 15979412
- [Background] Frank AM, Weidner T, Brynza J, Uckert W, Buchholz CJ, Hartmann J. CD8-Specific Designed Ankyrin Repeat Proteins Improve Selective Gene Delivery into Human and Primate T Lymphocytes. Hum Gene Ther. 2020 Jun;31(11-12):679-691. doi: 10.1089/hum.2019.248. Epub 2020 Apr 23. PMID 32160795
- [Background] Vormittag P, Gunn R, Ghorashian S, Veraitch FS. A guide to manufacturing CAR T cell therapies. Curr Opin Biotechnol. 2018 Oct;53:164-181. doi: 10.1016/j.copbio.2018.01.025. Epub 2018 Feb 18. PMID 29462761
- [Background] Zhou Q, Schneider IC, Edes I, Honegger A, Bach P, Schonfeld K, Schambach A, Wels WS, Kneissl S, Uckert W, Buchholz CJ. T-cell receptor gene transfer exclusively to human CD8(+) cells enhances tumor cell killing. Blood. 2012 Nov 22;120(22):4334-42. doi: 10.1182/blood-2012-02-412973. Epub 2012 Aug 16. PMID 22898597
- [Background] Smith TT, Stephan SB, Moffett HF, McKnight LE, Ji W, Reiman D, Bonagofski E, Wohlfahrt ME, Pillai SPS, Stephan MT. In situ programming of leukaemia-specific T cells using synthetic DNA nanocarriers. Nat Nanotechnol. 2017 Aug;12(8):813-820. doi: 10.1038/nnano.2017.57. Epub 2017 Apr 17. PMID 28416815
- [Background] Koneru M, Purdon TJ, Spriggs D, Koneru S, Brentjens RJ. IL-12 secreting tumor-targeted chimeric antigen receptor T cells eradicate ovarian tumors in vivo. Oncoimmunology. 2015 Jan 23;4(3):e994446. doi: 10.4161/2162402X.2014.994446. eCollection 2015 Mar. PMID 25949921
- [Background] Locke FL, Neelapu SS, Bartlett NL, Siddiqi T, Chavez JC, Hosing CM, Ghobadi A, Budde LE, Bot A, Rossi JM, Jiang Y, Xue AX, Elias M, Aycock J, Wiezorek J, Go WY. Phase 1 Results of ZUMA-1: A Multicenter Study of KTE-C19 Anti-CD19 CAR T Cell Therapy in Refractory Aggressive Lymphoma. Mol Ther. 2017 Jan 4;25(1):285-295. doi: 10.1016/j.ymthe.2016.10.020. Epub 2017 Jan 4. PMID 28129122
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- [Background] Neelapu SS, Tummala S, Kebriaei P, Wierda W, Gutierrez C, Locke FL, Komanduri KV, Lin Y, Jain N, Daver N, Westin J, Gulbis AM, Loghin ME, de Groot JF, Adkins S, Davis SE, Rezvani K, Hwu P, Shpall EJ. Chimeric antigen receptor T-cell therapy - assessment and management of toxicities. Nat Rev Clin Oncol. 2018 Jan;15(1):47-62. doi: 10.1038/nrclinonc.2017.148. Epub 2017 Sep 19. PMID 28925994